CLINICAL TRIAL: NCT00945204
Title: Evaluation of Intermediate Care Clinics for Diabetes
Acronym: ICCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals, Leicester (Other)
Collaborators: Warwick Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ICCD/NIHR SDO
Record Dates: First submitted 2009-07-23; First posted 2009-07-24 (Estimated); Last update posted 2012-08-08 (Estimated); Status verified 2012-08

CONDITIONS: Type 2 Diabetes
Keywords: type 2 diabetes; intermediate care; primary care; randomised controlled trial
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- access to intermediate care clinics (Experimental)
  Interventions: Other: intermediate care clinics (ICCs)
- usual care (No Intervention)

INTERVENTIONS:
Other: intermediate care clinics (ICCs) — The ICCs will be community based. Their aim is to support primary care, particularly smaller practices that have the most difficulty achieving good control. They will comprise a multidisciplinary team, and be led by specialist nurses who will place an emphasis on education and self management. Medical care will be provided by a diabetologist. The ICC will work closely with hospital based specialist teams and community services including podiatry and dietetics. Team members will work to local guidelines, adapted from national evidence based guidelines. Guidelines for referral to the ICCs will be common across all sites, and will include people with poorly controlled type 2 diabetes and those with poorly controlled cardiovascular risk factors.
  Arms: access to intermediate care clinics

SUMMARY:
The aim of this trial is to assess the effectiveness of intermediate care clinics for diabetes, compared to usual care.

DETAILED DESCRIPTION:
Intermediate care clinics (ICC) are suggested as one method of improving care for people with type 2 diabetes, but their effectiveness and cost effectiveness is not known. Their aim is to provide a multidisciplinary community based service to support general practices in achieving good control of their patients. Two local PCTs (Leicester City and Warwickshire) have agreed to establish intermediate care clinics as part of a cluster randomised trial of their effectiveness.

Patients with type 2 diabetes in participating practices will be invited to take part. Those that agree will attend a baseline assessment by a study nurse. This will include measurement of HbA1C, body mass index, waist circumference, blood pressure, urine and lipids, as well as questionnaires about quality of life, satisfaction with current services and continuity of care. Practices will then be randomised to either usual care or intervention arms, the latter having access to the new clinics. Participating patients will be asked to attend a follow up assessment 18-24 months after the baseline assessments, when the same measurements will be repeated. We expect about 30% of patients in the intervention arm will have been referred to the ICC.

The primary outcome will be the percentage of patients achieving adequate control of HbA1, blood pressure and cholesterol, comparing all participants in the intervention and control arms, whether or not those in the intervention arm attended ICC. The study is powered to detect a 10% difference in this outcome, and will include 51 practices and 5100 patients. We will also examine the effect of the intervention on process measures, such as the number of contacts in hospital and general practice. In the intervention arm we will document in detail the inputs provided by ICC, so that if successful the model can be adopted elsewhere.

The economic evaluation will be undertaken from a societal perspective. A costing study will measure intervention and treatment costs in both groups. A comparative assessment of the marginal costs and outcomes of the intervention will be undertaken, to include cost-effectiveness ratios and cost-utility analysis. All findings will be subject to sensitivity analysis.

Additionally we will explore the views of patients in the intervention arm who attended ICC using semi-structures interviews to identify positive and negative aspects of the patients' experiences. We will also hold focus groups to explore views of professional stakeholders.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes from participating practices across NHS Leicester, Warwickshire and Coventry.

Exclusion Criteria:

* Patients unable to give informed consent,
* Terminal cancer, OR
* Pregnant.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1997 (Actual)
Dates: Start 2007-05; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
The percentage of participants reaching target control of HbA1c (7.0), and blood pressure (<140/80) and cholesterol (<4 mmol/l), | 18 months

SECONDARY OUTCOMES:
Percentage of participants reaching target for individual risk factors (blood pressure, HbA1c or cholesterol) | 18 months
10 year risk for CHD and stroke assessed by the UKPDS risk engine | 18 months
Control of risk factors in all patients with type 2 diabetes in participating practices using anonymised routine data | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D Wilson, MD, Principal Investigator — University of Leicester
Locations (1):
- University of Leicester, Leicester, Leicestershire, United Kingdom

REFERENCES:
- [Derived] Wilson A, O'Hare JP, Hardy A, Raymond N, Szczepura A, Crossman R, Baines D, Khunti K, Kumar S, Saravanan P; ICCD trial group. Evaluation of the clinical and cost effectiveness of intermediate care clinics for diabetes (ICCD): a multicentre cluster randomised controlled trial. PLoS One. 2014 Apr 15;9(4):e93964. doi: 10.1371/journal.pone.0093964. eCollection 2014. PMID 24736243
- [Derived] Armstrong N, Baines D, Baker R, Crossman R, Davies M, Hardy A, Khunti K, Kumar S, O'Hare JP, Raymond N, Saravanan P, Stallard N, Szczepura A, Wilson A; ICCD Study Group. A cluster randomized controlled trial of the effectiveness and cost-effectiveness of intermediate care clinics for diabetes (ICCD): study protocol for a randomized controlled trial. Trials. 2012 Sep 12;13:164. doi: 10.1186/1745-6215-13-164. PMID 22971356